CLINICAL TRIAL: NCT06176092
Title: UCF Deciding Brains
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00005797
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Trust
Keywords: Healthy; Psychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Younger Adults (ages 20-39): The study will examine age differences in learning to trust using laboratory tasks and surveys.
- Older Adults (60 and older): The study will examine age differences in learning to trust using laboratory tasks and surveys.

SUMMARY:
The purpose of this research study is to understand how people make trust-related decisions in healthy aging.

Participants will be asked to complete one study session on the University of Central Florida (UCF) campus. The study session will be conducted in a private testing room and include a series of computerized cognitive tasks and learning games, as well as surveys of your beliefs, preferences, and past experiences.

The study will take a total of approximately 3.5 hours to completed. You will be allowed to take breaks during the session as needed. If you begin the study but do not complete the session, you will receive credit commensurate with your participation.

DETAILED DESCRIPTION:
Much of human interaction is based on trust. Optimal trust-related decision making and avoiding exploitation require the ability to learn about the trustworthiness of social partners across multiple interactions, but the role that learning plays in determining age deficits in trust decisions is currently unknown. To address this gap, this project will characterize basic cognitive processes in learning to trust and distrust in healthy aging.

The present study will examine age differences in learning to trust using laboratory tasks and surveys. The investigators hypothesize that social cues of trustworthiness will bias learning more in older adults (social cue bias, H1). Further, we predict that social cues of trustworthiness will interact with weighting of negative (loss aversion bias, H2) and recent (recency bias; H3) outcomes, and that these biases are exacerbated in older adults compared with younger adults (H4).

Young adult participants (age 20-39 years) will be recruited through the SONA pool. Older adult participants (age 60 and older) will be recruited from the University of Central Florida (UCF) Learning and Longevity Research Network (LLRN) registry and will be contacted by lab personnel via emails. Emails retrieved from the LLRN registry are provided by older-aged participants who wished to be contacted for research. Older adults will be screened to exclude those with cognitive impairment before being invited to participate. Those who meet criteria for inclusion in the study, will be scheduled for a study session in the lab.

ELIGIBILITY:
Inclusion Criteria:

* Younger adults only: Age 20-39 years old
* Older adults only: Age 60 years old and older
* Fluent English speaker
* At least 8th grade education
* On a stable regimen of medications
* Able to provide verbal and written informed consent
* Normal cognitive function

  * Older adults only: The above will be assessed/confirmed via cognitive screening assessments
  * Telephone Interview for Cognitive Status (TICS-M; see "Telephone Interview for Cognitive Status" in Local Site Documents)

Exclusion Criteria:

* Pregnant
* Presence of:

  * Schizophrenia Spectrum or Other Psychotic Disorders
  * Bipolar and Related Disorders
  * Depressive Disorders
  * Anxiety Disorders
  * Trauma- and Stressor-Related Disorders
  * Substance-Related and Addictive Disorders
* Current anticonvulsant, neuroleptic, or sedative use
* Uncorrected visual and hearing impairments
* Neurologic condition or event affecting the brain in the last 12 months (e.g., stroke, epilepsy, traumatic brain injury with >30-minute loss of consciousness)
* History of brain surgery including tumor resection, deep brain resection, pallidotomy, and thalamotomy
* Unstable medical illness (e.g., metastatic cancer)
* Significant cardiovascular condition or event in the last 12 months (e.g., major heart attack, heart bypass surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will target any healthy participants who are either between the ages of 20-39 or 60 and older.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
NIH Cognitive Toolbox | 1 year
  The NIH Toolbox which includes cognitive tasks to measure: Cognitive Function Composite Score, Fluid Cognition Composite Score, and Crystallized Cognition Composite Score
social Iowa Gambling Task (sIGT) | 1 year
  To investigate how older adults learn to trust others over multiple interactions, we developed the social Iowa Gambling Task (sIGT); modeled after the original Iowa Gambling Task.
Florida-Arizona Gambling Task (FLAG) | 1 year
  To examine choices between a sure offer and a draw from a deck of cards.
Phishing Email Suspicion Test (PEST) | 1 year
  This measures an individual's ability to detect phishing emails and has ecological validity pertaining to real-life internet fraud susceptibility.
Detection of Liars and Truth Tellers (LIE Task) | 1 year
  Participants will view brief videos of real crime suspects, who were either lying (liars) or telling the truth (truth tellers) about their involvement in the disappearance of a relative
Charity Task | 1 year
  This charity task assesses factors that can potentially influence charitable giving to organizations among younger and older adults, including familiarity, transparency, and personal importance.
Survey battery | 1 year
  The following surveys will that assess individual differences in CISDA factors and other potential exploitation risk predictors will be administered:
  (i) Theory of mind: (ii) Memory systems (iii) Socio-emotional processing (iv) Pain measures (v) Phishing vulnerability (vi) Demographics

CONTACTS AND LOCATIONS:
Overall Officials: Nichole Lighthall, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States